CLINICAL TRIAL: NCT02301702
Title: Evaluation of Tdap in Pregnancy to Prevent Infant Pertussis
Brief Title: Maternal Tdap Immunization in Guatemala
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Universidad del Valle, Guatemala (Other)
Responsible Party: Principal Investigator, Saad B. Omer, MBBS, MPH, PhD, Associate Professor of Global Health, Epidemiology, and Pediatrics, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00072201
Record Dates: First submitted 2014-11-22; First posted 2014-11-26 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Pertussis; Whooping Cough
Keywords: Maternal Immunization; Tdap; Td; Pertussis
MeSH Terms: conditions — Whooping Cough | interventions — Boostrix; adacel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tdap Vaccine (Experimental): Combination Tetnus Toxoid, Reduced Diptheria Toxoid and Acellular Pertusis (Tdap)
  Interventions: Biological: Tdap
- Td Vaccine (Active Comparator): Tetanus toxoid and reduced diphtheria toxoid vaccine (Td)
  Interventions: Biological: Td

INTERVENTIONS:
Biological: Tdap — Commercially available, U.S. and Guatemala licensed, 0.5mL intramuscular injection combination tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine
  Other Names: Boostrix, Adacel
  Arms: Tdap Vaccine
Biological: Td — The tetanus toxoid and reduced diphtheria toxoid vaccine (Td) used for this study will be the same preparation used by the National Immunization Program of Guatemala
  Arms: Td Vaccine

SUMMARY:
Maternal immunization with tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine (Tdap) is a potential strategy to protect young infants against pertussis before they are fully vaccinated because maternal antibodies may cross the placenta and passively protect her infant. The proposed study is a randomized, blinded, controlled, vaccine trial of maternal Tdap vaccination during the third trimester of pregnancy (Tdap vaccination at 27-36 weeks gestation). Pregnant women will be recruited from the prenatal care clinics at the Hospital Nacional Occidente and the Health Centers in Quetzaltenango, La Esperanza, San Juan Ostuncalco and Concepción Chiquirichapa. Enrolled women and their infants will be followed up until 7 months post-partum.

DETAILED DESCRIPTION:
The proposed study is a randomized, blinded, controlled, vaccine trial of maternal Tdap vaccination during the third trimester of pregnancy (Tdap vaccination at 27-36 weeks gestation). Pregnant women will be recruited from the prenatal care clinics at the Hospital Nacional de Occidente and the Health Centers in Quetzaltenango, La Esperanza, San Juan Ostuncalco and Concepción Chiquirichapa.

All healthy pregnant women between the ages of 18 and 40 years (inclusive) at 27 weeks gestation or later who are in the study areas will be eligible to participate in this study unless they meet one or more of the exclusion criteria. Pregnant women at <27 weeks gestation will be pre-screened and provided information about the study to encourage them to enroll later in their pregnancy. Women who are eligible will be enrolled after obtaining informed consent, and then they will be randomized to receive Tdap vaccine or Td vaccine. Enrolled women and their infants will be followed up until 7 months postpartum.

To address the primary objective, serum specimens will be collected from mothers prior to receiving the study product (Tdap or Td), within 72 hours after delivery and at 7 months post-partum. Moreover, infants specimens will be collected at delivery (cord blood or infant blood within 72 hours of birth), at 2 months of age (prior to the first dose of the routine childhood DTwP series), and at 7 months of age (approximately 4 weeks after the third dose of the routine DTwP series).

Infants will be given all three doses of the pentavalent vaccine which includes DTwP vaccine at 2, 4 and 6 months (routine childhood immunizations) as recommended by the immunization schedule of Guatemala's National Immunization Program.

Adverse events and serious adverse events will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman in late second or third trimester of pregnancy (i.e., after 27 weeks gestation),
2. Between the ages of 18 and 40 years (inclusive),
3. Intends to remain in the study area for at least seven months after delivery,
4. Has access to a mobile phone (defined as a phone in the possession of the participant or another family member with whom she lives),
5. Able to provide informed consent. If participant is illiterate, procedures to ensure full understanding of the research and consent process will be implemented according to international and federal guidelines.

Exclusion Criteria:

1. History of fever or oral temperature ≥ 38.0 degree Celsius within 48 hours prior to vaccination (women can be re-evaluated at a subsequent visit),
2. Received Tdap vaccine in the previous year,
3. History of serious systemic disease, including but not limited to: Guillain-Barré syndrome; known HIV, hepatitis B, or hepatitis C infection; heart/lung disease; uncontrolled diabetes mellitus (including gestational diabetes); chronic liver/kidney disease; clinically significant neurological disorders. This information will be based on self-reporting and (where possible) will be confirmed by health facility medical records.
4. High risk pregnancy, as identified by the Normas de Atención en Salud Integral, a guideline document published by the Ministry of Health, and also any previous complicated pregnancy or preterm delivery, spontaneous or medical abortion, or previous congenital anomaly,
5. Received immunoglobulin or other blood product within the preceding 3 month (with the exception of Rhogam),
6. History of allergy to any component of the vaccines (i.e. eggs, egg proteins, gelatin, formaldehyde, glutaraldehyde, polyethylene glycol p-isooctylphenyl ether, sucrose, aluminum hydroxide, polysorbate 80) or to latex,
7. History of severe reaction (including hypersensitivity) after receiving any vaccine,
8. History or evidence of immunosuppression (due to illness or treatment) or is on immunosuppressive therapy (includes long term use of steroids; use of high-dose inhaled steroids within past six months; with the exception of treatment with betamethasone or dexamethasone injections for the prevention of lung immaturity in the last trimester of pregnancy,
9. In the opinion of the study team - it would be unsafe or unsuitable for the pregnant mother or her fetus to receive the vaccine or participate in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 286 (Actual)
Dates: Start 2016-07; Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Infant pertussis antibody geometric mean concentrations (GMC) and 95% confidence intervals at birth (cord blood OR infant blood within 72 hours of birth), at 2 months of age, and 7 months of age | Birth to 7 months of age
Ratio of infant to mother pertussis antibody levels at the time of delivery | Birth to 7 months of age
Proportion of infants with at least a four-fold rise in serum antibody titer between 2 months and seven months of age (i.e., at four weeks after the 3rd dose of childhood DTwP) | Birth to 7 months of age
Maternal pertussis antibody GMC and 95% confidence intervals at baseline (pre-vaccination), within 72 hours after delivery, and seven months post-partum | Pre-vaccination to 7 months post-partum
Proportion of mothers sero-converting (serum pertussis antibody titer increase of ≥ 4-fold compared to pre-vaccination antibody levels) and 95% confidence intervals at the time of delivery (within 72 hours after delivery) and seven months post-partum | Pre-vaccination to 7 months post-partum

SECONDARY OUTCOMES:
Incidence of illnesses meeting the syndromic case definition (defined below); prematurity; pneumonia (per WHO Integrated Management of Childhood Illness [IMCI] classification) | Birth to 7 months of age
Birth weight and infant growth/anthropometric measurements (e.g., height and weight for age). | Birth to 7 months of age
Incidence of unsolicited non-serious (grades 1 & 2) adverse events 7 days post-delivery (for neonates) | Birth to 7 months of age
Infant growth/anthropometric measurements (e.g., height and weight z-scores at birth and 7 months of age) | Birth to 7 months of age
Incidence of serious (grades 3 & 4) adverse events through 7 months of age | Birth to 7 months of age
Laboratory (real-time PCR) confirmed pertussis infection in infants younger than 6 months of age | Birth to 7 months of age
Incidence of unsolicited non-serious (grades 1&2) AEs 28 days post vaccination | Pre-vaccination to 7 months post-partum
Incidence of serious (grades 3 & 4) adverse events through 7 months post-partum | Pre-vaccination to 7 months post-partum
Infant pertussis antibody geometric mean concentrations (GMC) and 95% confidence intervals at 19 months after delivery | Pre-vaccination to 19 mo post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Saad B. Omer, MBBS,MPH,PhD, Principal Investigator — Emory University
Locations (1):
- Universidad del Valle de Guatemala, Guatemala City, Guatemala